CLINICAL TRIAL: NCT06829446
Title: A Randomized Control Study of Repeat In-situ Ablation Versus Extensive Ablation for Patients with Recurrent Persistent Atrial Fibrillation
Brief Title: Recurrent Persistent Atrial Fibrillation:In-situ Ablation Vs Extensive Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Jinshan Hospital Affiliated to Fudan University (Unknown); Tongji University (Other)
Responsible Party: Principal Investigator, Xu Liu, Doctor Liu, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIEAF
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXT group (Experimental)
  Interventions: Procedure: Extra-PV extensive ablation; Procedure: Repeat same PVI and linear ablation as the first procedure
- IN-SITU group (Sham Comparator)
  Interventions: Procedure: Extra-PV extensive ablation; Procedure: Repeat same PVI and linear ablation as the first procedure

INTERVENTIONS:
Procedure: Extra-PV extensive ablation — Extra-PV extensive ablation
Procedure: Repeat same PVI and linear ablation as the first procedure — Repeat same PVI and linear ablation as the first procedure

SUMMARY:
This is an open label, randomized parallel control clinical trial, to compare extra-PV extensive ablation with in-situ ablation as two strategies for the treatment of PerAF to identify the mechanisms of PerAF recurrence.

DETAILED DESCRIPTION:
This is an open label, randomized parallel control clinical trial. Patients with recurrent persistent atrial fibrillation are 1:1 randomized into EXT group(Extra-PV extensive ablation) and IN-SITU group(Repeat same PVI and linear ablation as the first procedure). Postoperative recurrence rate and other indicators are analyzed to compare extra-PV extensive ablation with in-situ ablation as two strategies for the treatment of PerAF to identify the mechanisms of PerAF recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older; 2) Diagnosed as recurrent PerAF according to the latest clinical guidelines; 3) Ineffective or intolerable to ≥1 anti-arrhythmia drug treatment; 4) the first ablation procedure was PVI and linear ablation; 5) consented to receive radiofrequency catheter ablation.

Exclusion Criteria:

* 1) Recurrent atrial flutter/atrial tachycardia; 2) The first ablation procedure included extra-PV substrate ablation; 3) The first low voltage area>30%; 4) Serious complications during the first procedure; 5) The first ablation was paroxysmal atrial fibrillation. 6) Uncontrolled congestive heart failure; 7) History of severe valve disease and/or prosthetic valve replacement; 8) Left atrial thrombus confirmed by preoperative esophageal ultrasound; 9) Severe congenital heart disease; 10) Severe lung disease; 11) Left atrial diameter ≥60mm; 12) Contraindications for cardiac catheterization; 13) Myocardial infarction or stroke within 6 months; 14) Contrast agent allergy; 15) The use of anticoagulant drugs is contraindicated; 16) Have performed any cardiac surgery within 2 months;17) life expectancy is less than one year, including factors such as physical inability to tolerate ablation or unstable disease conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Freedom from any documented AF/AT episode | 12 months
  Freedom from any documented AF/AT episode lasting more than 30 seconds, excluding the initial 3 months blanking period, at a minimum of 12 months' follow-up after a single ablation procedure without antiarrhythmic medication.

SECONDARY OUTCOMES:
Freedom from any documented AF episode | 12 months
  Freedom from any documented AF episode lasting more than 30 seconds, excluding the initial 3 months blanking period, at a minimum of 12 months' follow-up after a single ablation procedure without antiarrhythmic medication
Any documented AT episode | 12 months
  Any documented AT episode lasting more than 30 seconds excluding the initial 3 months blanking period, at a minimum of 12 months' follow-up after a single ablation procedure without antiarrhythmic medication
Periprocedural complications | 12 months
  Periprocedural complications,including stroke, PV stenosis, cardiac perforation, oesophageal injury and death.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No